CLINICAL TRIAL: NCT00887289
Title: Non-interventional Observational Study on the Influence of Pramipexole (PPX) on Sensory Symptoms of Restless Legs Syndrome (RLS)
Brief Title: Non-interventional Observational Study on the Influence of Pramipexole on Sensory Symptoms of Restless Legs Syndrome (RLS)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.659
Record Dates: First submitted 2008-07-29; First posted 2009-04-23 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-03

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The main goal of this open-label, prospective, non-controlled, non-interventional post marketing surveillance study is to evaluate how pramipexole treatment works when applied in actual practice. In actual practice patients who would have been excluded in the clinical registration studies of pramipexole in moderate to severe primary Restless Legs Syndrome (i.e. those with certain disease histories, co-morbidities and/or demographic characteristics) will also be treated with pramipexole. Thus, during this post marketing surveillance study additional information on the efficacy and safety of pramipexole in those patients will be obtained. The objectives of this post marketing surveillance study are:

* To investigate the influence of Sifrol® (pramipexole) treatment on unpleasant sensory symptoms of Restless Legs Syndrome as measured with the short form of the McGill Pain Questionnaire.
* To assess if improvement of sensory symptoms correlates with overall Restless Legs Syndrome severity (International Restless Legs Syndrome Scale for Severity) and with secondary symptoms like sleeping problems and daytime tiredness (items 1 & 6 from Restless Legs Syndrome-6).
* To evaluate if the treatment effect of Sifrol on overall Restless Legs Syndrome severity (International Restless Legs Syndrome Scale for Severity) differs between patients with high pain scores and patients with lower pain scores.
* To compare General Practitioner and neurologist sites patient populations in terms of demographics, Restless Legs Syndrome severity at Visit 1 and treatment outcomes at Visit 3.
* To evaluate the development of behavioural changes under pramipexole treatment.

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of primary moderate to severe Restless Legs Syndrome.
2. Patients who are planned to be treated with Sifrol® (pramipexole) and where the decision of treatment is made independent of the patients' inclusion into this post marketing surveillance study.
3. Male or female patients aged at least 18 years.
4. Written informed consent by the patient for study participation.

Exclusion criteria:

1. Any contraindications according to the Summary of Product Characteristics: hypersensitivity to pramipexole or to any of the excipients.
2. Previous or ongoing treatment with Sifrol® (pramipexole).
3. Previous or ongoing treatment with dopamine receptor agonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RLS patients
Sampling Method: Non-Probability Sample
Enrollment: 1504 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (784):
- Germany (784):
  - Boehringer Ingelheim Investigational Site, Aalen
  - Boehringer Ingelheim Investigational Site 1, Achim
  - Boehringer Ingelheim Investigational Site 2, Achim
  - Boehringer Ingelheim Investigational Site 1, Ahrensburg
  - Boehringer Ingelheim Investigational Site 2, Ahrensburg
  - Boehringer Ingelheim Investigational Site, Albstadt
  - Boehringer Ingelheim Investigational Site, Alfeld
  - Boehringer Ingelheim Investigational Site, Allendorf
  - Boehringer Ingelheim Investigational Site 1, Alzenau in Unterfranken
  - Boehringer Ingelheim Investigational Site 2, Alzenau in Unterfranken
  - Boehringer Ingelheim Investigational Site, Anklam
  - Boehringer Ingelheim Investigational Site, Annaberg-Buchholz
  - Boehringer Ingelheim Investigational Site, Ansbach
  - Boehringer Ingelheim Investigational Site, Apolda
  - Boehringer Ingelheim Investigational Site, Arenshausen
  - Boehringer Ingelheim Investigational Site 1, Arnsberg
  - Boehringer Ingelheim Investigational Site 2, Arnsberg
  - Boehringer Ingelheim Investigational Site, Asperg
  - Boehringer Ingelheim Investigational Site 1, Attendorn
  - Boehringer Ingelheim Investigational Site 2, Attendorn
  - Boehringer Ingelheim Investigational Site, Aue
  - Boehringer Ingelheim Investigational Site 1, Augsburg
  - Boehringer Ingelheim Investigational Site 2, Augsburg
  - Boehringer Ingelheim Investigational Site 3, Augsburg
  - Boehringer Ingelheim Investigational Site, Aurich
  - Boehringer Ingelheim Investigational Site, Backnang
  - Boehringer Ingelheim Investigational Site, Bad Arolsen
  - Boehringer Ingelheim Investigational Site, Bad Bevensen
  - Boehringer Ingelheim Investigational Site, Bad Ems
  - Boehringer Ingelheim Investigational Site 1, Bad Hersfeld
  - Boehringer Ingelheim Investigational Site 2, Bad Hersfeld
  - Boehringer Ingelheim Investigational Site 1, Bad Honnef
  - Boehringer Ingelheim Investigational Site 2, Bad Honnef
  - Boehringer Ingelheim Investigational Site, Bad Krozingen
  - Boehringer Ingelheim Investigational Site, Bad Laer
  - Boehringer Ingelheim Investigational Site, Bad Lausick
  - Boehringer Ingelheim Investigational Site, Bad Marienberg
  - Boehringer Ingelheim Investigational Site 1, Bad Neuenahr-Ahrweiler
  - Boehringer Ingelheim Investigational Site 2, Bad Neuenahr-Ahrweiler
  - Boehringer Ingelheim Investigational Site, Bad Neustadt an der Saale
  - Boehringer Ingelheim Investigational Site, Bad Reichenhall
  - Boehringer Ingelheim Investigational Site, Bad Sachsa
  - Boehringer Ingelheim Investigational Site, Bad Salzuflen
  - Boehringer Ingelheim Investigational Site 1, Bad Salzungen
  - Boehringer Ingelheim Investigational Site 2, Bad Salzungen
  - Boehringer Ingelheim Investigational Site 3, Bad Salzungen
  - Boehringer Ingelheim Investigational Site, Bad Schwartau
  - Boehringer Ingelheim Investigational Site 1, Bad Segeberg
  - Boehringer Ingelheim Investigational Site 2, Bad Segeberg
  - Boehringer Ingelheim Investigational Site, Bad Sooden-Allendorf
  - Boehringer Ingelheim Investigational Site, Bad Tennstedt
  - Boehringer Ingelheim Investigational Site, Bad Wörishofen
  - Boehringer Ingelheim Investigational Site, Baden-Baden
  - Boehringer Ingelheim Investigational Site, Baesweiler
  - Boehringer Ingelheim Investigational Site 1, Bamberg
  - Boehringer Ingelheim Investigational Site 2, Bamberg
  - Boehringer Ingelheim Investigational Site 3, Bamberg
  - Boehringer Ingelheim Investigational Site, Baunatal
  - Boehringer Ingelheim Investigational Site, Bautzen
  - Boehringer Ingelheim Investigational Site 1, Bayreuth
  - Boehringer Ingelheim Investigational Site 2, Bayreuth
  - Boehringer Ingelheim Investigational Site, Bergheim
  - Boehringer Ingelheim Investigational Site 1, Bergkamen
  - Boehringer Ingelheim Investigational Site 2, Bergkamen
  - Boehringer Ingelheim Investigational Site 10, Berlin
  - Boehringer Ingelheim Investigational Site 11, Berlin
  - Boehringer Ingelheim Investigational Site 12, Berlin
  - Boehringer Ingelheim Investigational Site 13, Berlin
  - Boehringer Ingelheim Investigational Site 14, Berlin
  - Boehringer Ingelheim Investigational Site 15, Berlin
  - Boehringer Ingelheim Investigational Site 16, Berlin
  - Boehringer Ingelheim Investigational Site 17, Berlin
  - Boehringer Ingelheim Investigational Site 18, Berlin
  - Boehringer Ingelheim Investigational Site 19, Berlin
  - Boehringer Ingelheim Investigational Site 1, Berlin
  - Boehringer Ingelheim Investigational Site 20, Berlin
  - Boehringer Ingelheim Investigational Site 21, Berlin
  - Boehringer Ingelheim Investigational Site 22, Berlin
  - Boehringer Ingelheim Investigational Site 23, Berlin
  - Boehringer Ingelheim Investigational Site 24, Berlin
  - Boehringer Ingelheim Investigational Site 25, Berlin
  - Boehringer Ingelheim Investigational Site 26, Berlin
  - Boehringer Ingelheim Investigational Site 27, Berlin
  - Boehringer Ingelheim Investigational Site 28, Berlin
  - Boehringer Ingelheim Investigational Site 29, Berlin
  - Boehringer Ingelheim Investigational Site 2, Berlin
  - Boehringer Ingelheim Investigational Site 30, Berlin
  - Boehringer Ingelheim Investigational Site 31, Berlin
  - Boehringer Ingelheim Investigational Site 32, Berlin
  - Boehringer Ingelheim Investigational Site 33, Berlin
  - Boehringer Ingelheim Investigational Site 3, Berlin
  - Boehringer Ingelheim Investigational Site 4, Berlin
  - Boehringer Ingelheim Investigational Site 5, Berlin
  - Boehringer Ingelheim Investigational Site 6, Berlin
  - Boehringer Ingelheim Investigational Site 7, Berlin
  - Boehringer Ingelheim Investigational Site 8, Berlin
  - Boehringer Ingelheim Investigational Site 9, Berlin
  - Boehringer Ingelheim Investigational Site, Biberach
  - Boehringer Ingelheim Investigational Site, Bielefeld
  - Boehringer Ingelheim Investigational Site, Bingen
  - Boehringer Ingelheim Investigational Site, Bissendorf
  - Boehringer Ingelheim Investigational Site, Bitterfeld-Wolfen
  - Boehringer Ingelheim Investigational Site, Blankenhagen
  - Boehringer Ingelheim Investigational Site, Blaustein
  - Boehringer Ingelheim Investigational Site, Blieskastel
  - Boehringer Ingelheim Investigational Site 1, Bochum
  - Boehringer Ingelheim Investigational Site 2, Bochum
  - Boehringer Ingelheim Investigational Site 3, Bochum
  - Boehringer Ingelheim Investigational Site 4, Bochum
  - Boehringer Ingelheim Investigational Site 5, Bochum
  - Boehringer Ingelheim Investigational Site 6, Bochum
  - Boehringer Ingelheim Investigational Site 7, Bochum
  - Boehringer Ingelheim Investigational Site 1, Bockhorn
  - Boehringer Ingelheim Investigational Site 2, Bockhorn
  - Boehringer Ingelheim Investigational Site 1, Bodelshausen
  - Boehringer Ingelheim Investigational Site 2, Bodelshausen
  - Boehringer Ingelheim Investigational Site 1, Bonn
  - Boehringer Ingelheim Investigational Site 2, Bonn
  - Boehringer Ingelheim Investigational Site, Bordesholm
  - Boehringer Ingelheim Investigational Site, Bottrop
  - Boehringer Ingelheim Investigational Site, Braunschweig
  - Boehringer Ingelheim Investigational Site 1, Bremen
  - Boehringer Ingelheim Investigational Site 2, Bremen
  - Boehringer Ingelheim Investigational Site 3, Bremen
  - Boehringer Ingelheim Investigational Site 1, Bremerhaven
  - Boehringer Ingelheim Investigational Site 2, Bremerhaven
  - Boehringer Ingelheim Investigational Site 3, Bremerhaven
  - Boehringer Ingelheim Investigational Site, Breuberg
  - Boehringer Ingelheim Investigational Site, Bruchsal
  - Boehringer Ingelheim Investigational Site, Brühl
  - Boehringer Ingelheim Investigational Site, Buchbach
  - Boehringer Ingelheim Investigational Site, Burgdorf, Hanover
  - Boehringer Ingelheim Investigational Site, Burglengenfeld
  - Boehringer Ingelheim Investigational Site, Burscheid
  - Boehringer Ingelheim Investigational Site 1, Butzbach
  - Boehringer Ingelheim Investigational Site 2, Butzbach
  - Boehringer Ingelheim Investigational Site, Buxtehude
  - Boehringer Ingelheim Investigational Site, Büchen
  - Boehringer Ingelheim Investigational Site, Bückeburg
  - Boehringer Ingelheim Investigational Site, Calw
  - Boehringer Ingelheim Investigational Site 1, Celle
  - Boehringer Ingelheim Investigational Site 2, Celle
  - Boehringer Ingelheim Investigational Site 1, Chemnitz
  - Boehringer Ingelheim Investigational Site 2, Chemnitz
  - Boehringer Ingelheim Investigational Site 3, Chemnitz
  - Boehringer Ingelheim Investigational Site 4, Chemnitz
  - Boehringer Ingelheim Investigational Site 5, Chemnitz
  - Boehringer Ingelheim Investigational Site, Coburg
  - Boehringer Ingelheim Investigational Site, Coesfeld
  - Boehringer Ingelheim Investigational Site 1, Cologne
  - Boehringer Ingelheim Investigational Site 2, Cologne
  - Boehringer Ingelheim Investigational Site 3, Cologne
  - Boehringer Ingelheim Investigational Site 4, Cologne
  - Boehringer Ingelheim Investigational Site 5, Cologne
  - Boehringer Ingelheim Investigational Site 6, Cologne
  - Boehringer Ingelheim Investigational Site 7, Cologne
  - Boehringer Ingelheim Investigational Site 8, Cologne
  - Boehringer Ingelheim Investigational Site 9, Cologne
  - Boehringer Ingelheim Investigational Site, Cottbus
  - Boehringer Ingelheim Investigational Site 1, Crimmitschau
  - Boehringer Ingelheim Investigational Site 2, Crimmitschau
  - Boehringer Ingelheim Investigational Site, Dachau
  - Boehringer Ingelheim Investigational Site, Delbrück
  - Boehringer Ingelheim Investigational Site, Delmenhorst
  - Boehringer Ingelheim Investigational Site, Dernau
  - Boehringer Ingelheim Investigational Site 1, Dessau
  - Boehringer Ingelheim Investigational Site 2, Dessau
  - Boehringer Ingelheim Investigational Site 3, Dessau
  - Boehringer Ingelheim Investigational Site 4, Dessau
  - Boehringer Ingelheim Investigational Site 1, Dietzenbach
  - Boehringer Ingelheim Investigational Site 2, Dietzenbach
  - Boehringer Ingelheim Investigational Site 3, Dietzenbach
  - Boehringer Ingelheim Investigational Site, Dillingen
  - Boehringer Ingelheim Investigational Site, Dinkelsbühl
  - Boehringer Ingelheim Investigational Site 1, Dippoldiswalde
  - Boehringer Ingelheim Investigational Site 2, Dippoldiswalde
  - Boehringer Ingelheim Investigational Site 1, Dortmund
  - Boehringer Ingelheim Investigational Site 2, Dortmund
  - Boehringer Ingelheim Investigational Site 3, Dortmund
  - Boehringer Ingelheim Investigational Site 4, Dortmund
  - Boehringer Ingelheim Investigational Site, Döbeln
  - Boehringer Ingelheim Investigational Site 1, Dörentrup
  - Boehringer Ingelheim Investigational Site 2, Dörentrup
  - Boehringer Ingelheim Investigational Site 1, Dresden
  - Boehringer Ingelheim Investigational Site 2, Dresden
  - Boehringer Ingelheim Investigational Site 3, Dresden
  - Boehringer Ingelheim Investigational Site, Driedorf
  - Boehringer Ingelheim Investigational Site, Duderstadt
  - Boehringer Ingelheim Investigational Site 1, Duisburg
  - Boehringer Ingelheim Investigational Site 2, Duisburg
  - Boehringer Ingelheim Investigational Site 3, Duisburg
  - Boehringer Ingelheim Investigational Site, Durmersheim
  - Boehringer Ingelheim Investigational Site 1, Düsseldorf
  - Boehringer Ingelheim Investigational Site 2, Düsseldorf
  - Boehringer Ingelheim Investigational Site 3, Düsseldorf
  - Boehringer Ingelheim Investigational Site 4, Düsseldorf
  - Boehringer Ingelheim Investigational Site 5, Düsseldorf
  - Boehringer Ingelheim Investigational Site 6, Düsseldorf
  - Boehringer Ingelheim Investigational Site 7, Düsseldorf
  - Boehringer Ingelheim Investigational Site 8, Düsseldorf
  - Boehringer Ingelheim Investigational Site 9, Düsseldorf
  - Boehringer Ingelheim Investigational Site, Ebermannstadt
  - Boehringer Ingelheim Investigational Site 1, Edingen-Neckarhausen
  - Boehringer Ingelheim Investigational Site 2, Edingen-Neckarhausen
  - Boehringer Ingelheim Investigational Site, Edling
  - Boehringer Ingelheim Investigational Site, Eilenburg
  - Boehringer Ingelheim Investigational Site 1, Eisenach
  - Boehringer Ingelheim Investigational Site 2, Eisenach
  - Boehringer Ingelheim Investigational Site, Eisenberg
  - Boehringer Ingelheim Investigational Site, Eisenhüttenstadt
  - Boehringer Ingelheim Investigational Site, Ellwangen
  - Boehringer Ingelheim Investigational Site, Emmendingen
  - Boehringer Ingelheim Investigational Site, Emsdetten
  - Boehringer Ingelheim Investigational Site, Emskirchen
  - Boehringer Ingelheim Investigational Site, Enkirch
  - Boehringer Ingelheim Investigational Site, Ennigerloh
  - Boehringer Ingelheim Investigational Site, Eppelheim
  - Boehringer Ingelheim Investigational Site 1, Erbach im Odenwald
  - Boehringer Ingelheim Investigational Site 2, Erbach im Odenwald
  - Boehringer Ingelheim Investigational Site 3, Erbach im Odenwald
  - Boehringer Ingelheim Investigational Site 1, Erfurt
  - Boehringer Ingelheim Investigational Site 2, Erfurt
  - Boehringer Ingelheim Investigational Site 3, Erfurt
  - Boehringer Ingelheim Investigational Site, Erkrath
  - Boehringer Ingelheim Investigational Site 1, Erlangen
  - Boehringer Ingelheim Investigational Site, Eschborn
  - Boehringer Ingelheim Investigational Site, Eschlkam
  - Boehringer Ingelheim Investigational Site 10, Essen
  - Boehringer Ingelheim Investigational Site 11, Essen
  - Boehringer Ingelheim Investigational Site 12, Essen
  - Boehringer Ingelheim Investigational Site 13, Essen
  - Boehringer Ingelheim Investigational Site 14, Essen
  - Boehringer Ingelheim Investigational Site 1, Essen
  - Boehringer Ingelheim Investigational Site 2, Essen
  - Boehringer Ingelheim Investigational Site 3, Essen
  - Boehringer Ingelheim Investigational Site 4, Essen
  - Boehringer Ingelheim Investigational Site 5, Essen
  - Boehringer Ingelheim Investigational Site 6, Essen
  - Boehringer Ingelheim Investigational Site 7, Essen
  - Boehringer Ingelheim Investigational Site 8, Essen
  - Boehringer Ingelheim Investigational Site 9, Essen
  - Boehringer Ingelheim Investigational Site, Ettlingen
  - Boehringer Ingelheim Investigational Site, Extertal
  - Boehringer Ingelheim Investigational Site, Falkenhagen
  - Boehringer Ingelheim Investigational Site, Fehrbellin
  - Boehringer Ingelheim Investigational Site, Flintbek
  - Boehringer Ingelheim Investigational Site 1, Frankfurt
  - Boehringer Ingelheim Investigational Site 2, Frankfurt
  - Boehringer Ingelheim Investigational Site 3, Frankfurt
  - Boehringer Ingelheim Investigational Site, Freiberg
  - Boehringer Ingelheim Investigational Site 1, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 2, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 3, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 4, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 5, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site, Freilassing
  - Boehringer Ingelheim Investigational Site, Freinsheim
  - Boehringer Ingelheim Investigational Site 1, Freital
  - Boehringer Ingelheim Investigational Site 2, Freital
  - Boehringer Ingelheim Investigational Site 3, Freital
  - Boehringer Ingelheim Investigational Site, Friedrichshafen
  - Boehringer Ingelheim Investigational Site 1, Friedrichsthal
  - Boehringer Ingelheim Investigational Site 2, Friedrichsthal
  - Boehringer Ingelheim Investigational Site, Fulda
  - Boehringer Ingelheim Investigational Site, Fürstenfeldbruck
  - Boehringer Ingelheim Investigational Site 1, Fürstenwalde
  - Boehringer Ingelheim Investigational Site 2, Fürstenwalde
  - Boehringer Ingelheim Investigational Site, Fürstenzell
  - Boehringer Ingelheim Investigational Site 1, Fürth
  - Boehringer Ingelheim Investigational Site 2, Fürth
  - Boehringer Ingelheim Investigational Site, Gauting
  - Boehringer Ingelheim Investigational Site, Geisenhausen
  - Boehringer Ingelheim Investigational Site, Geithain
  - Boehringer Ingelheim Investigational Site 1, Gelnhausen
  - Boehringer Ingelheim Investigational Site 2, Gelnhausen
  - Boehringer Ingelheim Investigational Site 1, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 2, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 3, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 4, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site, Gera
  - Boehringer Ingelheim Investigational Site, Gerbstedt
  - Boehringer Ingelheim Investigational Site, Germering
  - Boehringer Ingelheim Investigational Site, Gersthofen
  - Boehringer Ingelheim Investigational Site, Giengen an der Brenz
  - Boehringer Ingelheim Investigational Site, Gladbeck
  - Boehringer Ingelheim Investigational Site, Gladenbach
  - Boehringer Ingelheim Investigational Site, Glauchau
  - Boehringer Ingelheim Investigational Site, Gleichen
  - Boehringer Ingelheim Investigational Site, Glienicke
  - Boehringer Ingelheim Investigational Site, Glücksburg
  - Boehringer Ingelheim Investigational Site, Gosheim
  - Boehringer Ingelheim Investigational Site, Göppingen
  - Boehringer Ingelheim Investigational Site 1, Göttingen
  - Boehringer Ingelheim Investigational Site 2, Göttingen
  - Boehringer Ingelheim Investigational Site 3, Göttingen
  - Boehringer Ingelheim Investigational Site 4, Göttingen
  - Boehringer Ingelheim Investigational Site 5, Göttingen
  - Boehringer Ingelheim Investigational Site, Gößweinstein
  - Boehringer Ingelheim Investigational Site, Greifswald
  - Boehringer Ingelheim Investigational Site, Greven
  - Boehringer Ingelheim Investigational Site, Grevenbroich
  - Boehringer Ingelheim Investigational Site, Großefehn
  - Boehringer Ingelheim Investigational Site, Großmaischeid
  - Boehringer Ingelheim Investigational Site 1, Grömitz
  - Boehringer Ingelheim Investigational Site 2, Grömitz
  - Boehringer Ingelheim Investigational Site, Grüna
  - Boehringer Ingelheim Investigational Site, Grünheide
  - Boehringer Ingelheim Investigational Site, Grünstadt
  - Boehringer Ingelheim Investigational Site, Gudensberg
  - Boehringer Ingelheim Investigational Site, Gundelfingen
  - Boehringer Ingelheim Investigational Site, Güster
  - Boehringer Ingelheim Investigational Site, Haag
  - Boehringer Ingelheim Investigational Site, Halbe
  - Boehringer Ingelheim Investigational Site 1, Halle
  - Boehringer Ingelheim Investigational Site 2, Halle
  - Boehringer Ingelheim Investigational Site 3, Halle
  - Boehringer Ingelheim Investigational Site 4, Halle
  - Boehringer Ingelheim Investigational Site 5, Halle
  - Boehringer Ingelheim Investigational Site 10, Hamburg
  - Boehringer Ingelheim Investigational Site 11, Hamburg
  - Boehringer Ingelheim Investigational Site 12, Hamburg
  - Boehringer Ingelheim Investigational Site 13, Hamburg
  - Boehringer Ingelheim Investigational Site 14, Hamburg
  - Boehringer Ingelheim Investigational Site 15, Hamburg
  - Boehringer Ingelheim Investigational Site 16, Hamburg
  - Boehringer Ingelheim Investigational Site 17, Hamburg
  - Boehringer Ingelheim Investigational Site 18, Hamburg
  - Boehringer Ingelheim Investigational Site 19, Hamburg
  - Boehringer Ingelheim Investigational Site 1, Hamburg
  - Boehringer Ingelheim Investigational Site 20, Hamburg
  - Boehringer Ingelheim Investigational Site 21, Hamburg
  - Boehringer Ingelheim Investigational Site 22, Hamburg
  - Boehringer Ingelheim Investigational Site 23, Hamburg
  - Boehringer Ingelheim Investigational Site 24, Hamburg
  - Boehringer Ingelheim Investigational Site 25, Hamburg
  - Boehringer Ingelheim Investigational Site 2, Hamburg
  - Boehringer Ingelheim Investigational Site 3, Hamburg
  - Boehringer Ingelheim Investigational Site 4, Hamburg
  - Boehringer Ingelheim Investigational Site 5, Hamburg
  - Boehringer Ingelheim Investigational Site 6, Hamburg
  - Boehringer Ingelheim Investigational Site 7, Hamburg
  - Boehringer Ingelheim Investigational Site 8, Hamburg
  - Boehringer Ingelheim Investigational Site 9, Hamburg
  - Boehringer Ingelheim Investigational Site, Hamelin
  - Boehringer Ingelheim Investigational Site, Hammelburg
  - Boehringer Ingelheim Investigational Site, Hamminkeln
  - Boehringer Ingelheim Investigational Site, Hannoversch Münden
  - Boehringer Ingelheim Investigational Site 1, Hanover
  - Boehringer Ingelheim Investigational Site 2, Hanover
  - Boehringer Ingelheim Investigational Site 3, Hanover
  - Boehringer Ingelheim Investigational Site 4, Hanover
  - Boehringer Ingelheim Investigational Site 5, Hanover
  - Boehringer Ingelheim Investigational Site 6, Hanover
  - Boehringer Ingelheim Investigational Site 7, Hanover
  - Boehringer Ingelheim Investigational Site 1, Harsewinkel
  - Boehringer Ingelheim Investigational Site 2, Harsewinkel
  - Boehringer Ingelheim Investigational Site 3, Harsewinkel
  - Boehringer Ingelheim Investigational Site, Hartenstein
  - Boehringer Ingelheim Investigational Site, Hasbergen
  - Boehringer Ingelheim Investigational Site, Heilbad Heiligenstadt
  - Boehringer Ingelheim Investigational Site 1, Heilbronn
  - Boehringer Ingelheim Investigational Site 2, Heilbronn
  - Boehringer Ingelheim Investigational Site 3, Heilbronn
  - Boehringer Ingelheim Investigational Site, Heinsberg
  - Boehringer Ingelheim Investigational Site, Herborn
  - Boehringer Ingelheim Investigational Site, Herbrechtingen
  - Boehringer Ingelheim Investigational Site, Herdorf
  - Boehringer Ingelheim Investigational Site, Herne
  - Boehringer Ingelheim Investigational Site, Herrenberg
  - Boehringer Ingelheim Investigational Site, Herrnhut
  - Boehringer Ingelheim Investigational Site, Herrsching am Ammersee
  - Boehringer Ingelheim Investigational Site 1, Herzogenrath
  - Boehringer Ingelheim Investigational Site 2, Herzogenrath
  - Boehringer Ingelheim Investigational Site, Hessisch Lichtenau
  - Boehringer Ingelheim Investigational Site, Hettstedt
  - Boehringer Ingelheim Investigational Site, Hildburghausen
  - Boehringer Ingelheim Investigational Site 1, Hildesheim
  - Boehringer Ingelheim Investigational Site 2, Hildesheim
  - Boehringer Ingelheim Investigational Site 3, Hildesheim
  - Boehringer Ingelheim Investigational Site 4, Hildesheim
  - Boehringer Ingelheim Investigational Site 1, Hof
  - Boehringer Ingelheim Investigational Site 2, Hof
  - Boehringer Ingelheim Investigational Site, Hohenprießnitz
  - Boehringer Ingelheim Investigational Site, Holle
  - Boehringer Ingelheim Investigational Site, Horb
  - Boehringer Ingelheim Investigational Site, Höchberg
  - Boehringer Ingelheim Investigational Site, Hückeswagen
  - Boehringer Ingelheim Investigational Site 1, Hüllhorst
  - Boehringer Ingelheim Investigational Site 2, Hüllhorst
  - Boehringer Ingelheim Investigational Site 3, Hüllhorst
  - Boehringer Ingelheim Investigational Site 1, Hürth
  - Boehringer Ingelheim Investigational Site 2, Hürth
  - Boehringer Ingelheim Investigational Site, Ibbenbueren
  - Boehringer Ingelheim Investigational Site 1, Ilmenau
  - Boehringer Ingelheim Investigational Site 2, Ilmenau
  - Boehringer Ingelheim Investigational Site, Immenstadt im Allgäu
  - Boehringer Ingelheim Investigational Site, Ingelfingen
  - Boehringer Ingelheim Investigational Site, Ingelheim
  - Boehringer Ingelheim Investigational Site, Ingolstadt
  - Boehringer Ingelheim Investigational Site, Inning am Ammersee
  - Boehringer Ingelheim Investigational Site, Irsch
  - Boehringer Ingelheim Investigational Site 1, Iserlohn
  - Boehringer Ingelheim Investigational Site 2, Iserlohn
  - Boehringer Ingelheim Investigational Site 1, Itzehoe
  - Boehringer Ingelheim Investigational Site 2, Itzehoe
  - Boehringer Ingelheim Investigational Site 3, Itzehoe
  - Boehringer Ingelheim Investigational Site, Jettingen
  - Boehringer Ingelheim Investigational Site 1, Jülich
  - Boehringer Ingelheim Investigational Site 2, Jülich
  - Boehringer Ingelheim Investigational Site 3, Jülich
  - Boehringer Ingelheim Investigational Site 1, Jüterbog
  - Boehringer Ingelheim Investigational Site 2, Jüterbog
  - Boehringer Ingelheim Investigational Site 1, Kaiserslautern
  - Boehringer Ingelheim Investigational Site 2, Kaiserslautern
  - Boehringer Ingelheim Investigational Site, Kamen
  - Boehringer Ingelheim Investigational Site, Kandel
  - Boehringer Ingelheim Investigational Site, Karlsfeld
  - Boehringer Ingelheim Investigational Site 1, Karlsruhe
  - Boehringer Ingelheim Investigational Site 2, Karlsruhe
  - Boehringer Ingelheim Investigational Site 1, Kassel
  - Boehringer Ingelheim Investigational Site 2, Kassel
  - Boehringer Ingelheim Investigational Site 3, Kassel
  - Boehringer Ingelheim Investigational Site 4, Kassel
  - Boehringer Ingelheim Investigational Site 1, Kaufbeuren
  - Boehringer Ingelheim Investigational Site 2, Kaufbeuren
  - Boehringer Ingelheim Investigational Site 3, Kaufbeuren
  - Boehringer Ingelheim Investigational Site 1, Kempten
  - Boehringer Ingelheim Investigational Site 2, Kempten
  - Boehringer Ingelheim Investigational Site, Kenzingen
  - Boehringer Ingelheim Investigational Site, Kernen
  - Boehringer Ingelheim Investigational Site, Kiel
  - Boehringer Ingelheim Investigational Site, Kirchardt
  - Boehringer Ingelheim Investigational Site, Kirchen
  - Boehringer Ingelheim Investigational Site, Kirchheim
  - Boehringer Ingelheim Investigational Site, Kirchheimbolanden
  - Boehringer Ingelheim Investigational Site, Kißlegg
  - Boehringer Ingelheim Investigational Site, Kleve
  - Boehringer Ingelheim Investigational Site, Klingenberg
  - Boehringer Ingelheim Investigational Site, Konz
  - Boehringer Ingelheim Investigational Site, Königsbrunn
  - Boehringer Ingelheim Investigational Site, Kösching
  - Boehringer Ingelheim Investigational Site, Köthen
  - Boehringer Ingelheim Investigational Site, Krefeld
  - Boehringer Ingelheim Investigational Site, Kreuztal
  - Boehringer Ingelheim Investigational Site, Kronach
  - Boehringer Ingelheim Investigational Site, Laage
  - Boehringer Ingelheim Investigational Site, Lahnau
  - Boehringer Ingelheim Investigational Site, Laichingen
  - Boehringer Ingelheim Investigational Site, Lampertheim
  - Boehringer Ingelheim Investigational Site, Landshut
  - Boehringer Ingelheim Investigational Site, Langen
  - Boehringer Ingelheim Investigational Site, Langerwehe
  - Boehringer Ingelheim Investigational Site, Lauterbach
  - Boehringer Ingelheim Investigational Site 1, Leipzig
  - Boehringer Ingelheim Investigational Site 2, Leipzig
  - Boehringer Ingelheim Investigational Site 3, Leipzig
  - Boehringer Ingelheim Investigational Site 4, Leipzig
  - Boehringer Ingelheim Investigational Site 5, Leipzig
  - Boehringer Ingelheim Investigational Site 6, Leipzig
  - Boehringer Ingelheim Investigational Site 7, Leipzig
  - Boehringer Ingelheim Investigational Site 8, Leipzig
  - Boehringer Ingelheim Investigational Site 9, Leipzig
  - Boehringer Ingelheim Investigational Site, Leverkusen
  - Boehringer Ingelheim Investigational Site, Lichtenfels
  - Boehringer Ingelheim Investigational Site 1, Limburg
  - Boehringer Ingelheim Investigational Site 2, Limburg
  - Boehringer Ingelheim Investigational Site 1, Limburgerhof
  - Boehringer Ingelheim Investigational Site 2, Limburgerhof
  - Boehringer Ingelheim Investigational Site, Lingen
  - Boehringer Ingelheim Investigational Site, Linz
  - Boehringer Ingelheim Investigational Site, Lippstadt
  - Boehringer Ingelheim Investigational Site, Lohr
  - Boehringer Ingelheim Investigational Site, Lubnjow
  - Boehringer Ingelheim Investigational Site, Ludwigsfelde
  - Boehringer Ingelheim Investigational Site 1, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 2, Ludwigshafen
  - Boehringer Ingelheim Investigational Site, Lübeck
  - Boehringer Ingelheim Investigational Site 1, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 2, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 1, Lüneburg
  - Boehringer Ingelheim Investigational Site 2, Lüneburg
  - Boehringer Ingelheim Investigational Site 1, Magdeburg
  - Boehringer Ingelheim Investigational Site 2, Magdeburg
  - Boehringer Ingelheim Investigational Site, Mainaschaff
  - Boehringer Ingelheim Investigational Site 1, Mannheim
  - Boehringer Ingelheim Investigational Site 2, Mannheim
  - Boehringer Ingelheim Investigational Site 3, Mannheim
  - Boehringer Ingelheim Investigational Site 4, Mannheim
  - Boehringer Ingelheim Investigational Site 5, Mannheim
  - Boehringer Ingelheim Investigational Site 6, Mannheim
  - Boehringer Ingelheim Investigational Site 7, Mannheim
  - Boehringer Ingelheim Investigational Site, Margetshöchheim
  - Boehringer Ingelheim Investigational Site, Markdorf
  - Boehringer Ingelheim Investigational Site, Markkleeberg
  - Boehringer Ingelheim Investigational Site 1, Marl
  - Boehringer Ingelheim Investigational Site 2, Marl
  - Boehringer Ingelheim Investigational Site, Mayen
  - Boehringer Ingelheim Investigational Site, Meckenheim
  - Boehringer Ingelheim Investigational Site, Meerbusch
  - Boehringer Ingelheim Investigational Site, Meinhard
  - Boehringer Ingelheim Investigational Site, Meißen
  - Boehringer Ingelheim Investigational Site, Mendig
  - Boehringer Ingelheim Investigational Site, Merseburg
  - Boehringer Ingelheim Investigational Site, Metzingen
  - Boehringer Ingelheim Investigational Site, Mittenwald
  - Boehringer Ingelheim Investigational Site, Mitterfelden
  - Boehringer Ingelheim Investigational Site, Molfsee
  - Boehringer Ingelheim Investigational Site, Monheim
  - Boehringer Ingelheim Investigational Site, Moormerland
  - Boehringer Ingelheim Investigational Site 1, Moosburg
  - Boehringer Ingelheim Investigational Site 2, Moosburg
  - Boehringer Ingelheim Investigational Site 1, Mosbach
  - Boehringer Ingelheim Investigational Site 2, Mosbach
  - Boehringer Ingelheim Investigational Site 1, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 2, Mönchengladbach
  - Boehringer Ingelheim Investigational Site, Murrhardt
  - Boehringer Ingelheim Investigational Site, Mutterstadt
  - Boehringer Ingelheim Investigational Site, Mühlheim
  - Boehringer Ingelheim Investigational Site, Mülheim
  - Boehringer Ingelheim Investigational Site 10, München
  - Boehringer Ingelheim Investigational Site 11, München
  - Boehringer Ingelheim Investigational Site 1, München
  - Boehringer Ingelheim Investigational Site 2, München
  - Boehringer Ingelheim Investigational Site 3, München
  - Boehringer Ingelheim Investigational Site 4, München
  - Boehringer Ingelheim Investigational Site 5, München
  - Boehringer Ingelheim Investigational Site 6, München
  - Boehringer Ingelheim Investigational Site 7, München
  - Boehringer Ingelheim Investigational Site 8, München
  - Boehringer Ingelheim Investigational Site 9, München
  - Boehringer Ingelheim Investigational Site, Münchweiler
  - Boehringer Ingelheim Investigational Site 1, Münster
  - Boehringer Ingelheim Investigational Site 2, Münster
  - Boehringer Ingelheim Investigational Site 3, Münster
  - Boehringer Ingelheim Investigational Site, Nagold
  - Boehringer Ingelheim Investigational Site, Naundorf
  - Boehringer Ingelheim Investigational Site, Nettetal
  - Boehringer Ingelheim Investigational Site 1, Neubrandenburg
  - Boehringer Ingelheim Investigational Site 2, Neubrandenburg
  - Boehringer Ingelheim Investigational Site, Neuhaus
  - Boehringer Ingelheim Investigational Site, Neuhof
  - Boehringer Ingelheim Investigational Site, Neukirchen-Vluyn
  - Boehringer Ingelheim Investigational Site, Neumarkt
  - Boehringer Ingelheim Investigational Site 1, Neuss
  - Boehringer Ingelheim Investigational Site 2, Neuss
  - Boehringer Ingelheim Investigational Site 3, Neuss
  - Boehringer Ingelheim Investigational Site 1, Neustadt
  - Boehringer Ingelheim Investigational Site 2, Neustadt
  - Boehringer Ingelheim Investigational Site 3, Neustadt
  - Boehringer Ingelheim Investigational Site, Neustrelitz
  - Boehringer Ingelheim Investigational Site, Niederlehme
  - Boehringer Ingelheim Investigational Site, Niedernwöhren
  - Boehringer Ingelheim Investigational Site, Nienstädt
  - Boehringer Ingelheim Investigational Site, Nordstemmen
  - Boehringer Ingelheim Investigational Site, Nossen
  - Boehringer Ingelheim Investigational Site, Notzingen
  - Boehringer Ingelheim Investigational Site 1, Nuremberg
  - Boehringer Ingelheim Investigational Site 2, Nuremberg
  - Boehringer Ingelheim Investigational Site 1, Oberhausen
  - Boehringer Ingelheim Investigational Site 2, Oberhausen
  - Boehringer Ingelheim Investigational Site 3, Oberhausen
  - Boehringer Ingelheim Investigational Site, Oberkirch
  - Boehringer Ingelheim Investigational Site, Oer-Erkenschwick
  - Boehringer Ingelheim Investigational Site, Offenbach
  - Boehringer Ingelheim Investigational Site, Offenburg
  - Boehringer Ingelheim Investigational Site, Olching
  - Boehringer Ingelheim Investigational Site 1, Oldenburg
  - Boehringer Ingelheim Investigational Site 2, Oldenburg
  - Boehringer Ingelheim Investigational Site, Olpe
  - Boehringer Ingelheim Investigational Site, Oppenheim
  - Boehringer Ingelheim Investigational Site, Oranienburg
  - Boehringer Ingelheim Investigational Site 1, Osnabrück
  - Boehringer Ingelheim Investigational Site 2, Osnabrück
  - Boehringer Ingelheim Investigational Site 3, Osnabrück
  - Boehringer Ingelheim Investigational Site 4, Osnabrück
  - Boehringer Ingelheim Investigational Site, Ostrach
  - Boehringer Ingelheim Investigational Site, Otterbach
  - Boehringer Ingelheim Investigational Site, Otterndorf
  - Boehringer Ingelheim Investigational Site, Ottobrunn bei München
  - Boehringer Ingelheim Investigational Site, Overath
  - Boehringer Ingelheim Investigational Site, Oy-Mittelberg
  - Boehringer Ingelheim Investigational Site 1, Paderborn
  - Boehringer Ingelheim Investigational Site 2, Paderborn
  - Boehringer Ingelheim Investigational Site 3, Paderborn
  - Boehringer Ingelheim Investigational Site 4, Paderborn
  - Boehringer Ingelheim Investigational Site 1, Parchim
  - Boehringer Ingelheim Investigational Site 2, Parchim
  - Boehringer Ingelheim Investigational Site, Parey
  - Boehringer Ingelheim Investigational Site, Passau
  - Boehringer Ingelheim Investigational Site 1, Peine
  - Boehringer Ingelheim Investigational Site 2, Peine
  - Boehringer Ingelheim Investigational Site, Peiting
  - Boehringer Ingelheim Investigational Site, Pfarrkirchen
  - Boehringer Ingelheim Investigational Site 1, Pforzheim
  - Boehringer Ingelheim Investigational Site 2, Pforzheim
  - Boehringer Ingelheim Investigational Site, Pirna
  - Boehringer Ingelheim Investigational Site, Plettenberg
  - Boehringer Ingelheim Investigational Site 1, Potsdam
  - Boehringer Ingelheim Investigational Site 2, Potsdam
  - Boehringer Ingelheim Investigational Site 3, Potsdam
  - Boehringer Ingelheim Investigational Site 4, Potsdam
  - Boehringer Ingelheim Investigational Site 5, Potsdam
  - Boehringer Ingelheim Investigational Site 6, Potsdam
  - Boehringer Ingelheim Investigational Site, Preetz
  - Boehringer Ingelheim Investigational Site, Prenzlau
  - Boehringer Ingelheim Investigational Site 1, Prien am Chiemsee
  - Boehringer Ingelheim Investigational Site 2, Prien am Chiemsee
  - Boehringer Ingelheim Investigational Site 1, Pulheim
  - Boehringer Ingelheim Investigational Site 2, Pulheim
  - Boehringer Ingelheim Investigational Site, Radeberg
  - Boehringer Ingelheim Investigational Site, Radevormwald
  - Boehringer Ingelheim Investigational Site, Rain
  - Boehringer Ingelheim Investigational Site 1, Rastatt
  - Boehringer Ingelheim Investigational Site, Regen
  - Boehringer Ingelheim Investigational Site 1, Regensburg
  - Boehringer Ingelheim Investigational Site 2, Regensburg
  - Boehringer Ingelheim Investigational Site 3, Regensburg
  - Boehringer Ingelheim Investigational Site 4, Regensburg
  - Boehringer Ingelheim Investigational Site, Reichenbach
  - Boehringer Ingelheim Investigational Site, Reinbek
  - Boehringer Ingelheim Investigational Site 1, Remscheid
  - Boehringer Ingelheim Investigational Site 2, Remscheid
  - Boehringer Ingelheim Investigational Site 3, Remscheid
  - Boehringer Ingelheim Investigational Site 4, Remscheid
  - Boehringer Ingelheim Investigational Site 5, Remscheid
  - Boehringer Ingelheim Investigational Site 6, Remscheid
  - Boehringer Ingelheim Investigational Site, Rendsburg
  - Boehringer Ingelheim Investigational Site, Rheine
  - Boehringer Ingelheim Investigational Site, Rodewisch
  - Boehringer Ingelheim Investigational Site 1, Rostock
  - Boehringer Ingelheim Investigational Site 2, Rostock
  - Boehringer Ingelheim Investigational Site 3, Rostock
  - Boehringer Ingelheim Investigational Site 4, Rostock
  - Boehringer Ingelheim Investigational Site, Röcknitz
  - Boehringer Ingelheim Investigational Site, Rödermark
  - Boehringer Ingelheim Investigational Site, Rüsselsheim am Main
  - Boehringer Ingelheim Investigational Site, Saarbrücken
  - Boehringer Ingelheim Investigational Site, Salzgitter
  - Boehringer Ingelheim Investigational Site, Scharnebeck
  - Boehringer Ingelheim Investigational Site, Schirgiswalde
  - Boehringer Ingelheim Investigational Site, Schleching
  - Boehringer Ingelheim Investigational Site, Schleiden
  - Boehringer Ingelheim Investigational Site, Schleswig
  - Boehringer Ingelheim Investigational Site, Schloß Holte-Stukenbrock
  - Boehringer Ingelheim Investigational Site, Schönebeck
  - Boehringer Ingelheim Investigational Site, Schönfeld
  - Boehringer Ingelheim Investigational Site, Schriesheim
  - Boehringer Ingelheim Investigational Site, Schwaig
  - Boehringer Ingelheim Investigational Site, Schwalmstadt
  - Boehringer Ingelheim Investigational Site, Schwanewede
  - Boehringer Ingelheim Investigational Site, Schwarzenbach A Wald
  - Boehringer Ingelheim Investigational Site, Schwarzenberg
  - Boehringer Ingelheim Investigational Site, Schwarzenbruck
  - Boehringer Ingelheim Investigational Site 1, Schwäbisch Gmünd
  - Boehringer Ingelheim Investigational Site 2, Schwäbisch Gmünd
  - Boehringer Ingelheim Investigational Site, Schwerte
  - Boehringer Ingelheim Investigational Site, Seeheim-Jugenheim
  - Boehringer Ingelheim Investigational Site, Seifhennersdorf
  - Boehringer Ingelheim Investigational Site, Selbitz
  - Boehringer Ingelheim Investigational Site, Senden
  - Boehringer Ingelheim Investigational Site, Sendenhorst
  - Boehringer Ingelheim Investigational Site, Senftenberg
  - Boehringer Ingelheim Investigational Site, Siegen
  - Boehringer Ingelheim Investigational Site, Sigmaringen
  - Boehringer Ingelheim Investigational Site, Simmern
  - Boehringer Ingelheim Investigational Site, Sindelfingen
  - Boehringer Ingelheim Investigational Site, Sinsheim
  - Boehringer Ingelheim Investigational Site, Soest
  - Boehringer Ingelheim Investigational Site 1, Sondershausen
  - Boehringer Ingelheim Investigational Site 2, Sondershausen
  - Boehringer Ingelheim Investigational Site, Sonsbeck
  - Boehringer Ingelheim Investigational Site 1, Sömmerda
  - Boehringer Ingelheim Investigational Site 2, Sömmerda
  - Boehringer Ingelheim Investigational Site, Spremberg
  - Boehringer Ingelheim Investigational Site 1, Stade
  - Boehringer Ingelheim Investigational Site 2, Stade
  - Boehringer Ingelheim Investigational Site, Stamsried
  - Boehringer Ingelheim Investigational Site, Steinfeld
  - Boehringer Ingelheim Investigational Site, Steinmauern
  - Boehringer Ingelheim Investigational Site, Stendal
  - Boehringer Ingelheim Investigational Site, Sternberg
  - Boehringer Ingelheim Investigational Site, Stolberg
  - Boehringer Ingelheim Investigational Site, Stollberg
  - Boehringer Ingelheim Investigational Site, Stolpen
  - Boehringer Ingelheim Investigational Site, Stotternheim
  - Boehringer Ingelheim Investigational Site, Straelen
  - Boehringer Ingelheim Investigational Site, Stralsund
  - Boehringer Ingelheim Investigational Site, Straubing
  - Boehringer Ingelheim Investigational Site, Stuhr
  - Boehringer Ingelheim Investigational Site 10, Stuttgart
  - Boehringer Ingelheim Investigational Site 11, Stuttgart
  - Boehringer Ingelheim Investigational Site 1, Stuttgart
  - Boehringer Ingelheim Investigational Site 2, Stuttgart
  - Boehringer Ingelheim Investigational Site 3, Stuttgart
  - Boehringer Ingelheim Investigational Site 4, Stuttgart
  - Boehringer Ingelheim Investigational Site 5, Stuttgart
  - Boehringer Ingelheim Investigational Site 6, Stuttgart
  - Boehringer Ingelheim Investigational Site 7, Stuttgart
  - Boehringer Ingelheim Investigational Site 8, Stuttgart
  - Boehringer Ingelheim Investigational Site 9, Stuttgart
  - Boehringer Ingelheim Investigational Site, Telgte
  - Boehringer Ingelheim Investigational Site, Templin
  - Boehringer Ingelheim Investigational Site, Tirschenreuth
  - Boehringer Ingelheim Investigational Site 1, Trier
  - Boehringer Ingelheim Investigational Site 2, Trier
  - Boehringer Ingelheim Investigational Site 3, Trier
  - Boehringer Ingelheim Investigational Site, Ulm
  - Boehringer Ingelheim Investigational Site, Übach-Palenberg
  - Boehringer Ingelheim Investigational Site 1, Velen
  - Boehringer Ingelheim Investigational Site 2, Velen
  - Boehringer Ingelheim Investigational Site, Vellmar
  - Boehringer Ingelheim Investigational Site, Velten
  - Boehringer Ingelheim Investigational Site, Verden an der Aller
  - Boehringer Ingelheim Investigational Site, Viersen
  - Boehringer Ingelheim Investigational Site 1, Vilshofen
  - Boehringer Ingelheim Investigational Site 2, Vilshofen
  - Boehringer Ingelheim Investigational Site 3, Vilshofen
  - Boehringer Ingelheim Investigational Site, Visselhövede
  - Boehringer Ingelheim Investigational Site, Waghäusel
  - Boehringer Ingelheim Investigational Site, Wahlstedt
  - Boehringer Ingelheim Investigational Site, Wald-Michelbach
  - Boehringer Ingelheim Investigational Site, Waldkraiburg
  - Boehringer Ingelheim Investigational Site, Wandlitz
  - Boehringer Ingelheim Investigational Site, Wankendorf
  - Boehringer Ingelheim Investigational Site, Warthausen
  - Boehringer Ingelheim Investigational Site, Wegberg
  - Boehringer Ingelheim Investigational Site, Wehrsdorf
  - Boehringer Ingelheim Investigational Site, Weingarten
  - Boehringer Ingelheim Investigational Site, Weinsberg
  - Boehringer Ingelheim Investigational Site, Weißenfels
  - Boehringer Ingelheim Investigational Site, Welbsleben
  - Boehringer Ingelheim Investigational Site, Welver
  - Boehringer Ingelheim Investigational Site, Wernigerode
  - Boehringer Ingelheim Investigational Site, Werningshausen
  - Boehringer Ingelheim Investigational Site, Wesel
  - Boehringer Ingelheim Investigational Site, Wessobrunn
  - Boehringer Ingelheim Investigational Site 1, Westoverledingen
  - Boehringer Ingelheim Investigational Site 2, Westoverledingen
  - Boehringer Ingelheim Investigational Site 1, Wiesbaden
  - Boehringer Ingelheim Investigational Site 2, Wiesbaden
  - Boehringer Ingelheim Investigational Site 3, Wiesbaden
  - Boehringer Ingelheim Investigational Site, Wiesenfelden
  - Boehringer Ingelheim Investigational Site, Wietzen
  - Boehringer Ingelheim Investigational Site, Wildau
  - Boehringer Ingelheim Investigational Site, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site, Wilhermsdorf
  - Boehringer Ingelheim Investigational Site, Willich
  - Boehringer Ingelheim Investigational Site, Winkelhaid
  - Boehringer Ingelheim Investigational Site, Winsen
  - Boehringer Ingelheim Investigational Site 1, Wismar
  - Boehringer Ingelheim Investigational Site 2, Wismar
  - Boehringer Ingelheim Investigational Site 3, Wismar
  - Boehringer Ingelheim Investigational Site, Wissen
  - Boehringer Ingelheim Investigational Site, Wittgensdorf
  - Boehringer Ingelheim Investigational Site 1, Witzenhausen
  - Boehringer Ingelheim Investigational Site 2, Witzenhausen
  - Boehringer Ingelheim Investigational Site 3, Witzenhausen
  - Boehringer Ingelheim Investigational Site, Wolfenbüttel
  - Boehringer Ingelheim Investigational Site 1, Wolfratshausen
  - Boehringer Ingelheim Investigational Site 2, Wolfratshausen
  - Boehringer Ingelheim Investigational Site 3, Wolfratshausen
  - Boehringer Ingelheim Investigational Site, Wolfsburg
  - Boehringer Ingelheim Investigational Site 1, Wolgast
  - Boehringer Ingelheim Investigational Site, Worms
  - Boehringer Ingelheim Investigational Site, Wörrstadt
  - Boehringer Ingelheim Investigational Site 1, Wörth
  - Boehringer Ingelheim Investigational Site 2, Wörth
  - Boehringer Ingelheim Investigational Site, Wunstorf
  - Boehringer Ingelheim Investigational Site 1, Wuppertal
  - Boehringer Ingelheim Investigational Site 2, Wuppertal
  - Boehringer Ingelheim Investigational Site 3, Wuppertal
  - Boehringer Ingelheim Investigational Site 4, Wuppertal
  - Boehringer Ingelheim Investigational Site, Wustrau
  - Boehringer Ingelheim Investigational Site, Würzburg
  - Boehringer Ingelheim Investigational Site, Zeitz
  - Boehringer Ingelheim Investigational Site, Zella-Mehlis
  - Boehringer Ingelheim Investigational Site, Zerbst
  - Boehringer Ingelheim Investigational Site, Ziltendorf
  - Boehringer Ingelheim Investigational Site, Zirndorf
  - Boehringer Ingelheim Investigational Site, Zorge
  - Boehringer Ingelheim Investigational Site, Zschopau
  - Boehringer Ingelheim Investigational Site 1, Zwickau
  - Boehringer Ingelheim Investigational Site 2, Zwickau
  - Boehringer Ingelheim Investigational Site, Zwönitz

RESULTS

PARTICIPANT FLOW:
Groups:
- Pramipexole: 0.088 mg every day (qd), titration up to 0.54 mg qd possible
Period: Overall Study
Arm/Group | Pramipexole
Started | 1504
Completed | 1409
Not Completed | 95
Not completed — Lack of Efficacy | 14
Not completed — Adverse Event | 27
Not completed — Withdrawal by Subject | 26
Not completed — Lost to Follow-up | 8
Not completed — Other | 20

BASELINE CHARACTERISTICS:
Arm/Group | Pramipexole
Number analyzed (Participants) | 1504
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (13.0)
Gender [Number; unit: participants]
  Female | 1008
  Male | 490

OUTCOME MEASURES:

1. Primary Outcome: Summary of Change From Baseline in Total Sum of McGill Pain Questionnaire to Visit 3
Description: Change in Total Sum Score of McGill Pain Questionnaire at Visit 3 to baseline. The sum scores can have values in the range from 0 (no pain) to 20 (worst pain). A negative change is an improvement of pain, a positive change a worsening of pain.
Time Frame: Baseline to Visit 3
Population: Full analysis set, no imputation technique was applied
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 1320
Scores on scale | -14.48 (9.69)

2. Primary Outcome: Summary of Change From Baseline in Total Sum of McGill Pain Questionnaire to Visit 3 for Patients Treated by General Practitioner
Description: as for outcome 1
Time Frame: Baseline to Visit 3
Population: All patients of the full analysis set treated by a general practitioner, no imputation technique was applied
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 830
Scores on scale | -15.87 (9.39)

3. Primary Outcome: Summary of Change From Baseline in Total Sum of McGill Pain Questionnaire to Visit 3 for Patients Treated by Neurologist
Description: as for outcome 1
Time Frame: Baseline to Visit 3
Population: All patients of the full analysis set treated by a neurologist, no imputation technique was applied
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 490
Scores on scale | -12.13 (9.73)

4. Secondary Outcome: Summary of Change From Baseline in Restless Legs Syndrome Severity Scale With 6 Questions to Visit 3
Description: Change in RLS-6 at Visit 3 to baseline. The sum scores can have values in the range from 0 (best) to 20 (worst) A negative change is an improvement of RLS-6, a positive change a worsening of RLS-6.
Time Frame: Baseline to Visit 3
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 1391
Scores on scale | -1.63 (0.98)

5. Secondary Outcome: Summary of Change From Baseline in International Restless Legs Syndrome Scale for Severity to Visit 3
Description: Change in IRLS at Visit 3 to baseline. The sum scores can have values in the range from 0 (best) to 40 (worst) A negative change is an improvement of IRLS, a positive change a worsening of IRLS.
Time Frame: Baseline to Visit 3
Population: Full analysis set, no imputation technique was applied
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 1364
Scores on scale | -17.71 (8.86)

6. Secondary Outcome: Behavioural Changes During Treatment
Description: Number of patients with occurence of behavioural changes in terms of impulse control disorders
Time Frame: Baseline to Visit 3
Population: Full analysis set, no imputation technique was applied
Measure: Number; unit: participants
Arm/Group | Pramipexole
Number analyzed (Participants) | 1492
participants | 8

ADVERSE EVENTS:
Time Frame: 14 Weeks
Arm/Group | Pramipexole
Serious Adverse Events (participants affected / at risk) | 6/1504
Other Adverse Events (participants affected / at risk) | 0/1504
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole (N=1504)
Death (General disorders) | 2
Muscoloskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gallbladder operation (Surgical and medical procedures) | 1
Hospitalization (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.